CLINICAL TRIAL: NCT03489460
Title: Research Exploring Sleep Education & Technology
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-01591
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Sleep Health
Keywords: sleep health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive sleep health messages + GAD (Active Comparator): Procedures will be delivered to users of the GAD, individuals who have opted in via their smartphone application, to receive messages about various areas of health.
  Interventions: Behavioral: Specialized sleep-related message interventions; Behavioral: GAD
- Sleep message No GAD (Active Comparator): For two weeks participants agree to receive sleep health messages and wear the GAD
  Interventions: Behavioral: Specialized sleep-related message interventions

INTERVENTIONS:
Behavioral: Specialized sleep-related message interventions — Over the course of 2 weeks' participants will receive specialized sleep-related message interventions to encourage sleep awareness via the smartphone application.
Behavioral: GAD — Survey responses will be merged with objective GAD data (sleep time, time in deep sleep, physical activity) which will assist in developing message design formats for message testing.
  Arms: Receive sleep health messages + GAD

SUMMARY:
A pilot study that seeks to develop a set of typologies of users of mobile sleep tracking technologies, and optimal sleep health educational strategies among users of mobile wearable technologies that track sleep.

ELIGIBILITY:
Inclusion Criteria:

* A current user of the OURA ring activity and sleep tracker device.

For Aim 3 MOST message testing, the inclusion criteria include the following:

* Health conscious.

Exclusion Criteria:

* Non English speakers.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Sleep time measured by wearable mobile sleep tracking technology | 15 Days
  Mobile sleep tracking device will be worn by patient for 15 days and will measure sleep patterns in patients
Time in deep sleep measured by wearable mobile sleep tracking technology | 15 Days
  Mobile sleep tracking device will be worn by patient for 15 days and will measure sleep patterns in patients
Dysfunctional Beliefs about Sleep (DBAS) scale | 1 Day
  24-item DBAS scale with five subscales corresponding to: (1) consequences of insomnia (2) control and predictability of sleep (3) sleep requirement expectations (5) sleep-promoting practices
Measure of motivation to change using the Change Assessment Scale (CAS) | 15 Days
  8 scale measure divided into 4 separate scales: Scale 1: "Pre-Contemplation" Scale 2: "Contemplation" Scale 3 "Action" Scale 4 "Maintenance"

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: Requests should be directed to Rebecca.robbins@nyulangone.org. To gain access, data requestors will need to sign a data access agreement